CLINICAL TRIAL: NCT07100132
Title: Research on the Clinical Value of Cranial CT and CTA in Patients With Cerebral Hemorrhage
Brief Title: Research on the Clinical Value of Cranial CT and CTA for Cerebral Hemorrhage Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GE2023JZ-01
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Intracerebral Hemorrhage (ICH)
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Based on the patients' neurological functional outcomes, they were categorized into a good prognosis

SUMMARY:
The objective of this observational study is to investigate the predictive value of various imaging signs in patients with intracerebral hemorrhage, thereby providing a reference for clinical diagnosis and treatment. The primary aim is to evaluate the association between specific imaging signs and both hematoma expansion and poor outcomes in these patients.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients who were confirmed to have cerebral hemorrhage through head CT imaging examination upon admission; (2) Those who completed head CT and CTA within 8 hours of onset and had a follow-up CT within 24 hours of admission; (3) With complete clinical data.

Exclusion Criteria:

(1) Patients who cannot complete CT and CTA within the prescribed time; (2) Patients with secondary cerebral hemorrhage due to cerebral vascular malformations, brain tumors, brain trauma, cerebral aneurysms, etc.; (3) Patients who have been taking oral anticoagulants for a long time or have blood system diseases; (4) Primary intraventricular hemorrhage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebral hemorrhage treated at the Affiliated Hospital of Guizhou Medical University
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Randomized 180-day mRS score of 0-3 (%) | From the end of the six-month period after discharge.

IPD SHARING:
Plan to Share IPD: Yes